CLINICAL TRIAL: NCT03244514
Title: Biomarker-guided Implementation of the Cardiovascular (CV) Surgery AKI Bundle to Reduce the Occurrence of AKI After Cardiac Surgery- Prevention of AKI
Brief Title: Biomarker-guided Implementation of the AKI Bundle
Acronym: PrevAKI-mc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: European Society of Intensive Care Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 07-AnIt-16
Record Dates: First submitted 2017-07-07; First posted 2017-08-09 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Acute Kidney Injury (Nontraumatic)
Keywords: cardiac surgery; KDIGO-Guideline
MeSH Terms: conditions — Acute Kidney Injury | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Implementation of the cardiovascular surgery AKI bundle
  1. discontinuation of all nephrotoxic agents when possible
  2. optimization of volume status and hemodynamic parameters
  3. close monitoring of serum creatinine, fluid balance and urinary output
  4. avoidance of hyperglycemia
  5. considerations of alternatives to radiocontrast agents
  6. discontinuation of angiotensin converting enzyme inhibitors and angiotensin receptor blockers in the perioperative period
  7. avoidance of HES, gelatin, and chlorid-rich solutions
  Interventions: Other: Intervention
- Control group (No Intervention): The patients will receive standard of care (according to each center)

INTERVENTIONS:
Other: Intervention — Implementation of the cardiovascular AKI bundle (see arm description)
  Arms: Intervention group

SUMMARY:
There is no specific therapy for acute kidney injury. It is presumed that supportive measures improve the care and outcome of patients with acute kidney injury.

The investigators hypothesize that the implementation of a bundle of supportive measures adapted to patients undergoing cardiovascular surgery reduces the occurence of AKI.

A Randomized prospective multicenter trial is needed to investigate whether the implementation of the bundle of measures is effective to prevent AKI in high risk patients undergoing cardiac surgery. In this feasibility trial the investigators will analyze the compliance rate to the trial protocol in a multicenter, multinational cohort in preparation for a large randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac surgery with cardiopulmonary bypass (CPB)
* Urinary [TIMP-2] * [IGFBP7] >= 0.3 4h after CPB
* Written informed consent

Exclusion Criteria:

* Preexisting AKI (stage 1 and higher)
* Patients with cardiac assist devices (ECMO, LVAD, RVAD, IABP)
* Pregnancy, breastfeeding
* Known (Glomerulo-)-Nephritis, intersstitial nephritis or vasculitis
* CKD with eGFR < 20 mL/min
* Dialyses dependent CKD
* Prior kidney transplant within the last 12 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2019-10-26 (Actual); Study Completion 2020-01-26 (Actual)

PRIMARY OUTCOMES:
Compliance rate | 48 hours after start of intervention
  proportion of patients who are treated according to the trial protocol: CV surgery AKI bundle fulfilled at all time

SECONDARY OUTCOMES:
Occurence of AKI | 72 hours after start of intervention
Moderate and severe AKI | 72 hours after start of intervention
Free-days through of vasoactive medications and mechanical ventilation | 28 days after start of intervention
Renal recovery | 90 days after start of intervention
  renal recovery is defined as serum creatinine levels < 0.5 mg/dl higher than baseline serum creatinine (creatinine level before surgery)
Mortality | 90 days after start of intervention
ICU and hospital stay | up to 1 year after start of intervention (until discharge)
Number of patients with renal replacement therapy | 90 days after start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Zarbock, PhD, Study Chair — University Hospital Muenster, Dept. of Anesthesiology
Locations (12):
- Belgium (3):
  - CHU Brugmann, Intensive Care Medicine, Brussels
  - AZ Maria Middelares, Ghent
  - Universitair Ziekenhuis Gent, Ghent
- Germany (4):
  - Universitätsklinikum Bergmannsheil Bochum, Bochum
  - Universitätsklinikum Gießen, Klinik für Herz-, Kinderherz- und Gefäßchirurgie, Giessen
  - Philipps-Universität Marburg, Marburg
  - University Hospital Muenster, Münster
- Italy (2):
  - Ospedale San Raffaele S.r.I., I.R.C.C.S., Milan
  - Centro Cardiologico Monzino Istituto di Ricovero e Cura a Carattere Scientific, Milan
- Hospital del la Santa Creu i Sant Pau; Unidad de Cuidados Intensivos, Barcelona, Spain
- United Kingdom (2):
  - St. Thomas' Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meersch M, Schmidt C, Hoffmeier A, Van Aken H, Wempe C, Gerss J, Zarbock A. Prevention of cardiac surgery-associated AKI by implementing the KDIGO guidelines in high risk patients identified by biomarkers: the PrevAKI randomized controlled trial. Intensive Care Med. 2017 Nov;43(11):1551-1561. doi: 10.1007/s00134-016-4670-3. Epub 2017 Jan 21. PMID 28110412
- [Derived] Zarbock A, Kullmar M, Ostermann M, Lucchese G, Baig K, Cennamo A, Rajani R, McCorkell S, Arndt C, Wulf H, Irqsusi M, Monaco F, Di Prima AL, Garcia Alvarez M, Italiano S, Miralles Bagan J, Kunst G, Nair S, L'Acqua C, Hoste E, Vandenberghe W, Honore PM, Kellum JA, Forni LG, Grieshaber P, Massoth C, Weiss R, Gerss J, Wempe C, Meersch M. Prevention of Cardiac Surgery-Associated Acute Kidney Injury by Implementing the KDIGO Guidelines in High-Risk Patients Identified by Biomarkers: The PrevAKI-Multicenter Randomized Controlled Trial. Anesth Analg. 2021 Aug 1;133(2):292-302. doi: 10.1213/ANE.0000000000005458. PMID 33684086
- [Derived] Kullmar M, Massoth C, Ostermann M, Campos S, Grau Novellas N, Thomson G, Haffner M, Arndt C, Wulf H, Irqsusi M, Monaco F, Di Prima A, Garcia Alvarez M, Italiano S, Cegarra SanMartin V, Kunst G, Nair S, L'Acqua C, Hoste EAJ, Vandenberghe W, Honore PM, Kellum J, Forni L, Grieshaber P, Weiss R, Gerss J, Wempe C, Meersch M, Zarbock A. Biomarker-guided implementation of the KDIGO guidelines to reduce the occurrence of acute kidney injury in patients after cardiac surgery (PrevAKI-multicentre): protocol for a multicentre, observational study followed by randomised controlled feasibility trial. BMJ Open. 2020 Apr 6;10(4):e034201. doi: 10.1136/bmjopen-2019-034201. PMID 32265240